CLINICAL TRIAL: NCT00502567
Title: A Phase 1, Open Label Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2171 and Selected Chemotherapy Regimens When Given in Combination to Patients With Advanced Solid Tumors
Brief Title: A Study to Assess Safety, Tolerability and PK of AZD2171 and Chemotherapy on Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00008
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumors; AZD2171; Phase I
MeSH Terms: interventions — cediranib; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Pemetrexed; Irinotecan; Cetuximab; Docetaxel

INTERVENTIONS:
Drug: AZD2171 — oral tablet once daily
  Other Names: cediranib; RECENTIN™.
Drug: FOLFOX — intravenous infusion
  Other Names: 5-Fluorouracil, Leucovorin and Oxaliplatin
Drug: Pemetrexed — intravenous infusion
  Other Names: Alimta®; Pemetrexed disodium
Drug: Irinotecan (administered with & without Cetuximab) — intravenous injection
  Other Names: Campto®; Camptosar®; irinotecan hydrochloride
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere®

SUMMARY:
A multicentre, 2-part study to assess the safety and tolerability of once daily oral doses of AZD2171 when administered with various anticancer regimens (part A) and to confirm the tolerability of its combination with FOLFOX (part B).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed metastatic cancer that is not amenable to surgery or radiation therapy with curative intent
* measurable lesion by CT or other techniques according to RECIST

Exclusion Criteria:

* Inadequate bone marrow reserve
* history of poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-01; Primary Completion 2007-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of once daily oral doses of AZD2171 when given in combination with one of these anticancer regimens; FOLFOX, Pemetrexed, Irinotecan, Docetaxel | After 5 weeks of treatment

SECONDARY OUTCOMES:
Examine the PK interaction of AZD2171 with one of the 4 different chemotherapeutic regimens. Make a preliminary evaluation of clinical response as measured by objective response rate. | Assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca; Bijoyesh Mookerjee, MD, Study Chair — AstraZeneca; Patricia LoRusso, DO, Principal Investigator — Wayne State University
Locations (3):
- United States (3):
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Nashville, Tennessee